CLINICAL TRIAL: NCT06965556
Title: A Prospective Study to Evaluate the Clinical Significance of Medical Humanities-based Patient Education Strategy for Breast Cancer Patients During Perioperative Hospitalization Stage
Brief Title: Patient Education Strategy for Breast Cancer Patients During Perioperative Hospitalization Stage
Acronym: PE-CAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE-CAT
Record Dates: First submitted 2025-04-16; First posted 2025-05-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Patient Education; Perioperative Care; Psychological Intervention
Keywords: breast carcinoma; patient education; educational comic; psychological intervention; hospitalization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Humanities-based Patient Education Strategy (Active Comparator): Mental Enhanced Education Strategy
  Patients allocated to the enhanced mental health education intervention cohort will receive supplemental medical humanities modules alongside the standard Practical Education Strategy during hospitalization. This content is derived from a comic publication compiled by the breast surgery team of Fudan University Shanghai Cancer Center, which narrates the 4600-year human battle against breast cancer in a grand story. The content combines humorous cartoons with novel-like text, covering the evolution of human understanding of breast cancer, and the emergence and development of various therapies, drugs, and technologies. For patients unable to read, audio books and dynamic cartoon videos are available on mobile devices. The general content framework is as follows:
  * Understanding of breast cancer in ancient Egypt and Persia;
  * Hippocratic-Galenic Theories: early management of breast disorders in Greco-Roman antiquity;
  * Traditional Chinese medical interpret
  Interventions: Other: Medical Humanities-based Patient Education Strategy
- Routine Patient Education Strategy (No Intervention): Practical Education Strategy
  Admission Day
  * Comprehensive admission nursing assessment and introduction to care protocols: Admission assessment form, nutritional assessment, fall risk assessment, deep vein thrombosis risk assessment, pain assessment, etc.
  * Orientation to ward environment and policies: introduction to the medical team, online doctor-patient communication platform, ward facilities, daily routines, dietary guidelines, and other essential services, etc.
  * Review of medical history and guidance on preoperative examinations and precautions: Hematological tests, electrocardiogram, ultrasound, mammography, CT, MRI, core needle biopsy, fine needle aspiration, etc.
  Days Before Surgery
  * Personal preparation instructions: Bathing, hair washing, fasting, and fluid restriction guidelines, etc.
  * Interpretation of preoperative examination results.
  * Overview of common surgical approaches for breast cancer, introduction of surgery options based on the condition, especially emphasis on

INTERVENTIONS:
Other: Medical Humanities-based Patient Education Strategy — Medical Humanities-based Patient Education with Comic-based Medical Education Materials for Breast Cancer Patients during Perioperative Hospitalization Stage
  Arms: Medical Humanities-based Patient Education Strategy

SUMMARY:
Introduction Breast cancer remains a leading global health concern, with significant psychological challenges during the perioperative period. Traditional patient education focuses on disease management but often neglects emotional and cognitive needs. Perioperative inpatients are relatively stable and have the time and mental space for deeper education and psychological support. This study evaluates the clinical significance of a medical humanities-based education strategy for breast cancer patients during hospitalization, aiming to enhance psychological resilience, treatment adherence, and quality of life.

Methods and Analysis This prospective, non-randomized, open-label study will include female patients with early-stage breast cancer scheduled for surgery at Fudan University Shanghai Cancer Center. Participants will be allocated to two cohorts: practical education group and mental enhanced group. The primary endpoint is psychological assessment at hospital discharge, including anxiety (GAD-7), depression (PHQ-9), and sleep quality (ISI). Secondary endpoints include the proportion of patients opting for breast-conserving procedures, incidence of postoperative complications, long-term treatment adherence (MMAS-8), patients' disease-coping resilience (CD-RISC-10), and quality of life assessment (EORTC QLQ instruments) at 12-month follow-up. Data collection and statistical analysis will be conducted using validated instruments and software, with significance set at p ≤0.05.

Ethics and Dissemination Approved by the FUSCC ethics committee, all participants provide informed consent. Results will be disseminated through international conferences and peer-reviewed journals. The study adheres to ethical guidelines, ensuring data confidentiality via encrypted platforms. Authors declare no conflicts of interest, supported by Shanghai Municipal Science and Technology Innovation Action Plan (24DZ2303500). Findings aim to optimize perioperative education strategies, addressing psychological and informational needs of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Female
* Patient with early-stage breast cancer with preoperative pathology confirming invasive breast carcinoma or ductal carcinoma in situ
* No clinical or imaging evidence of distant metastasis
* Patients to receive breast surgery during hospitalizaiton (including mastectomy, breast conserving therapy, reconstrucion, etc.)
* Be able and willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

* Patients with locally advanced breast cancer to receive neoadjuvant therapy
* Patients currently participating in other clinical trials, which may have impact on the participation in this trial
* Previous history of breast cancer (patients with ipsilateral recurrence after breast sparing surgery)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1138 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
anxiety status at hospital discharge | Five days after surgery
  anxiety status at hospital discharge evaluated using the GAD-7 questionnaire Generalized Anxiety Disorder scale, GAD-7 (0-21 points): Cut-off values of 5, 10, and 15 delineated mild, moderate, and severe anxiety
depression severity at hospital discharge | Five days after surgery
  depression severity at hospital discharge assessed with the PHQ-9 instrument Patient Health Questionnaire, PHQ-9 (0-27 points): Thresholds at 5, 10, 15, and 20 classified mild, moderate, moderately severe, and severe depression.
sleep quality at hospital discharge | Five days after surgery
  sleep quality at hospital discharge measured via the ISI scale Insomnia Severity Index, ISI (0-28 points): Scores ≥8, ≥15, and ≥22 indicated subthreshold, moderate, and severe insomnia.

SECONDARY OUTCOMES:
The proportion of patients opting for breast-conserving cosmetic procedures | Five days after surgery
  including breast-conserving surgery, oncoplastic breast-conserving surgery, implant-based or autologous breast reconstruction
Incidence of postoperative complications requiring surgical intervention | 12 months follow-up
  Incidence of postoperative complications requiring surgical intervention within 12 months after surgery
Long-term treatment adherence | 12 months follow-up
  Long-term treatment adherence evaluation at the 12-month postoperative follow-up (assessed using the MMAS-8 scale) 8-item Morisky Medication Adherence Scale, MMAS-8 (0-8 points): Medication adherence was categorized as optimal (≥6) or suboptimal.
Patients' disease-coping resilience | 12 months follow-up
  Patients' disease-coping resilience at 12 months postoperatively (evaluated with the CD-RISC-10 instrument) (10-item Connor-Davidson Resilience Scale, CD-RISC-10 (0-40 points): Psychological resilience was dichotomized using the 29.5 threshold (high vs. low resilience).
Quality of life assessment at discharge | Five days after surgery
  Quality of life assessment (EORTC QLQ-BR23) at discharge EORTC QLQ instruments (BR23 breast-specific module): Quality-of-life metrics were standardized using European Organization for Research and Treatment of Cancer linear transformation protocols (0-100 scoring)
Quality of life assessment | 12 months follow-up
  Quality of life assessment (EORTC BR45) 1 year postoperatively EORTC QLQ instruments (BR45 comprehensive module): Quality-of-life metrics were standardized using European Organization for Research and Treatment of Cancer linear transformation protocols (0-100 scoring)
Loss to follow-up rate | 12 months follow-up
  Loss to follow-up rate between study groups at 12-month follow-up
Quality of life assessment | 12 months follow-up
  Quality of life assessment (EORTC QLQ-C30) 1 year postoperatively EORTC QLQ instruments (C30 core module): Quality-of-life metrics were standardized using European Organization for Research and Treatment of Cancer linear transformation protocols (0-100 scoring)
Quality of life assessment at discharge | Five days after surgery
  Quality of life assessment (EORTC QLQ-C30/BR45) at hospital discharge EORTC QLQ instruments (C30 core module): Quality-of-life metrics were standardized using European Organization for Research and Treatment of Cancer linear transformation protocols (0-100 scoring)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR